CLINICAL TRIAL: NCT03567200
Title: A League of Their Own: Examining the Effectiveness of a Psycho-social and Sport Program Targeting At-risk Adolescent Girls
Brief Title: Girls United on the Move: A Unique Integrated Physical Activity and Psychosocial Program for At-risk Adolescent Girls
Acronym: GUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Cristina Caperchione, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H17-01540
Record Dates: First submitted 2018-05-15; First posted 2018-06-25 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Chewing Gum; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-Arm Feasibility (Experimental): 9-week, 1x/week, 90-minute face-to-face sessions.
  Interventions: Behavioral: Single-Arm Feasibility

INTERVENTIONS:
Behavioral: Single-Arm Feasibility — Participants in each of the 8 participating groups (N=10-12 per group) are exposed to an integrated intervention program (integration of physical activity and psychosocial components). Each session is co-facilitated by a trained research staff member and a registered social worker, providing participants with the opportunity to engage in physical activity behaviours as well as discuss various psychosocial topics that are applicable to the participants interests. Physical activities include participating in group activities such as rock climbing, self-defence, yoga, etc. Psychosocial topics addressed include group discussions around cyber-bullying, sexual abuse and exploitation, gender issues, etc.
  Other Names: Girls United and On the Move (GUM) Intervention

SUMMARY:
The purpose of this project is to evaluate the effectiveness of a 9-week psycho-social and physical activity program aimed at improving body image, physical self-perceptions, and self-compassion for at-risk adolescent girls. In collaboration with the Elizabeth Fry Society, the GUM program will be delivered to at-risk adolescent girls within the Okanagan Region. Information will be gathered concerning program content and delivery, as well as insights into the participants' experiences with the program. These results will provide much needed information about whether programs integrating psychological, social, and physical components of health are beneficial for this population.

DETAILED DESCRIPTION:
Body dissatisfaction increases throughout adolescence; strong associations have been established between body image emotions and negative self--perceptions, reduced self-compassion, low self- esteem, and depression in adolescent girls. This is heightened in at--risk adolescent girls, including those of low socioeconomic status, who have experienced abuse and who have limited social support. As such, unique strategies aimed at reducing negative self--perceptions of one's physical self and improving self- compassion among at--risk adolescent girls are needed. Engagement in physical activity is one way in which adolescent girls may experience positive self--perceptions, enhanced body image emotions, and increased self--compassion, yet the research has primarily focused on girls who are already involved in organized physical activities (i.e., athletes). To address this need, the research team and representatives from the Central Okanagan Elizabeth Fry Society, a National charitable organisation dedicated to advancing the safety, legal rights, and economic security of women and children, have co--created the unique 9- week Girls United and on the Move (GUM) integrated program (psycho-social and physical activity) to improve physical self--perception, body image, and self--compassion among at--risk adolescent girls living in the Okanagan Region of British Columbia. This is particularly important in the Okanagan where there is a high number of adolescent girls from low income, abusive households, with many facing sexual exploitation and extreme despair, compared to other adolescent girls in British Columbia. Thus, the current aim is to implement and undertake a comprehensive evaluation of the program's effectiveness in terms of physical self--perceptions, body image, self--compassion, and commitment to and enjoyment of physical activity, in order to refine and deliver the program more widely.

This 9- week, integrated program will be implemented in up to 8 middle schools throughout the Okanagan. It includes a 1.5 hour, weekly session held at local schools and facilitated by a trained researcher and registered social worker. These sessions include psycho-social components (e.g., understanding healthy relationships, building self--confidence) in addition to engaging in various physical activities (e.g., soccer, dance, and martial arts). At--risk adolescent girls from the participating schools will be identified and recruited by school counsellors. Each school group will include 10- to 12 participants, yielding a total sample of approximately 80-100.

ELIGIBILITY:
Inclusion Criteria:

* Participants who identify with experiencing challenges with personal or family lives.
* Must identify as female between the ages of 11-15 years of age.

Exclusion Criteria:

* No specific exclusion criteria, however, only girls that are specifically identified and invited to join GUM by the school guidance counsellors, at the participating middle schools, will be invited to participate in the research.

Ages: 11 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 83 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Body Image | Assessing change from baseline to post-intervention (9-weeks).
  Measured using the Physical Self-Description Questionnaire (PSDQ), which is a multidimensional tool used to measure physical self--perceptions, body image and self--concept. The purpose of the PSDQ is to see how people describe themselves physically.
Self-Compassion | Assessing change from baseline to post-intervention (9-weeks).
  Measured using the Self-Compassion Scale (SCS), which is a a valid and reliable 26--item scale that has previously been used in this population.
Physical Self-Perceptions | Assessing change from baseline to post-intervention (9-weeks).
  Measured using the Physical Self-Description Questionnaire (PSDQ), which is a multidimensional tool used to measure physical self--perceptions, body image and self--concept. The purpose of the PSDQ is to see how people describe themselves physically.

SECONDARY OUTCOMES:
Sport Enjoyment and Commitment | Assessing change from baseline to post-intervention (9-weeks).
  Measured using the Sport-Commitment Questionnaire, which is a 58-item questionnaire that addresses five components or sub-scales which are believed to impact sport commitment; this includes sport enjoyment, involvement alternatives, personal investments, social constraints, and involvement opportunities. Not only has this construct been shown to be very important in motivating youth in sport, but it also may indicate the positive affect to commitment in youth sport programs.
Participant satisfaction and acceptability of the GUM program | Post-Intervention (9-weeks)
  Assessed by conducting semi-structured interviews to gather information concerning program content and delivery, as well as insights into their experiences with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Caperchione, PhD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Okanagan, Kelowna, British Columbia, Canada

REFERENCES:
- [Derived] Caperchione CM, Hargreaves N, Sabiston CM, Berg S, Kowalski KC, Ferguson LJ. Exploring the Effectiveness of an Integrated Physical Activity and Psychosocial Program Targeting At-Risk Adolescent Girls: Protocol for the Girls United and on the Move (GUM) Intervention Study. JMIR Res Protoc. 2020 Jun 9;9(6):e15302. doi: 10.2196/15302. PMID 32515748